CLINICAL TRIAL: NCT06483516
Title: Post-operative Quality of Life After AAA Management: EVAR Versus Open Repair
Status: Recruiting | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Clinical Professor, University Paul Sabatier of Toulouse
Other Study IDs: QOL AAA
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Quality of Life After AAA Surgery
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OPEN REPAIR: Patient operated for AAA by conventional surgery
  Interventions: Procedure: Open repair
- ENDO REPAIR: Patient operated for AAA by Endovascular exclusion (EVAR/F-BEVAR)
  Interventions: Procedure: Endovascular repair

INTERVENTIONS:
Procedure: Open repair — Open repair via median laparotomy or lumbotomy
  Groups: OPEN REPAIR
Procedure: Endovascular repair — EVAR if AAA simple F-BEVAR if Complex AAA
  Groups: ENDO REPAIR

SUMMARY:
The treatment of AAA has been revolutionised by minimally invasive techniques that allow patients to return home more quickly and have a reputation for having a low impact on their quality of life.

However, no study has looked at the quality of life of patients treated for AAA using open or endovascular surgery, using a scale adapted to post-operative follow-up.

The investigators conducted a single-centre prospective observational study to assess the quality of life of patients undergoing AAA surgery by endovascular exclusion or open surgery

DETAILED DESCRIPTION:
Aneurysms of the abdominal aorta are common in patients over the age of 65. Treatment methods to prevent rupture have changed considerably since the 2000s, with the advent of minimally invasive endovascular techniques. These minimally invasive techniques, which have the reputation of enabling patients to return home quickly without any loss of quality of life, have been called into question over time by the appearance of secondary endoleaks, leading to re-interventions and significant secondary ruptures.

Open aortic surgery is often described as invasive and burdensome for patients, with a lasting result in terms of efficacy in treating AAA, but at the cost of a major deterioration in patients' quality of life.

The literature presents numerous studies of postoperative quality of life, using general scales that have not been validated specifically for postoperative use. Furthermore, all these studies do not take into account the patient's pre-operative state and are therefore unable to provide an objective view of changes in quality of life and post-operative recovery after open surgery or evar. The QoR15 is a questionnaire comprising 15 questions specifically validated for the study of patients' early postoperative recovery.

In order to obtain objective data, the investigators conducted a single-centre prospective observational study to assess the quality of life of patients undergoing AAA surgery by endovascular exclusion or open surgery

ELIGIBILITY:
Inclusion Criteria:

* Aortic abdominal aneurysm above 50mm

Exclusion Criteria:

* Emergent surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient to be operated on for an aneurysm of the abdominal aorta in scheduled surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life evolution | Day before surgery/ the day of discharge home (up to 1 month) / 1 month after surgery post operative consultation/ 6 months after surgery post operative consultation
  Qor15 score filled by the patient

SECONDARY OUTCOMES:
Post operative mortality | day 30
  Death after surgery
early Reintervention | Day 30
  New operation
late reintervention | 3 months, 6 months, yearly
  New operation

CONTACTS AND LOCATIONS:
Locations (1):
- Hostalrich, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided